CLINICAL TRIAL: NCT02931760
Title: Placement Of Cardiac PacemaKer Trial (POCKET)-RCT
Acronym: POCKET-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Gävleborg (Other)
Responsible Party: Principal Investigator, Peter Magnusson, M.D., Cardiologist, Region Gävleborg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016371
Record Dates: First submitted 2016-10-01; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Pacemaker Ddd

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- subcutaneous pacemaker (Active Comparator): The patients who are randomized to receive a subcutaneously implanted pacemaker
  Interventions: Device: subcutaneous pacemaker
- intramuscular pacemaker (Active Comparator): The patients who are randomized to receive an intramuscular implanted pacemaker
  Interventions: Device: intramuscular pacemaker

INTERVENTIONS:
Device: subcutaneous pacemaker — During implant of a pacemaker the device is either implanted subcutaneously or intramuscular
  Arms: subcutaneous pacemaker
Device: intramuscular pacemaker — During implant of a pacemaker the device is either implanted subcutaneously or intramuscular
  Arms: intramuscular pacemaker

SUMMARY:
Aim: To compare patient satisfaction with intramuscular placement of a pacemaker pocket to subcutaneous placement.

Patients will be randomized (approximately half i each group) to receive the pacemaker device either subcutaneously (current practise) or intramuscular)

DETAILED DESCRIPTION:
Background: Implantation of a cardiac pacemaker may be indicated in patients with a significant bradycardia according to current guidelines.1 Annually, around 691 pacemakers per million inhabitants are implanted in Sweden.2 A pacemaker system consist of one or two leads connected to a device that is implanted beneath the collarbone.3,4 Vessel access is typically on the left side through the cephalic, axillary or subclavian vein. The pacemaker is inserted into a pocket. Routinely this pocket is just above the pectoral fascia (subcutaneously) or sometimes in skinny patients with a small amount of subcutaneous fat between the pectoral muscular layer (intramuscular). Even though technical developments have diminished the size of pacemakers markedly over time, complications due to superficial implants still do occur.5,6 Occasionally the device erode the skin and a complete extraction of the system is necessary. More frequently patients complain about the device being too superficial which sometimes require surgical repositioning of the device.5,6 The device may create discomfort, pain, and unsightly.5,6 The lateral corner of the device may disturb the shoulder movement, sleep and the leads can be turned within the pocket (Twiddler's syndrome). Minor branches from the supraclavicular nerves may result in discomfort. When vessels from the subcutaneous adipose tissue are distorted, extensive bruising may be bothersome and a large hematoma is a known risk of infection. The perfusion in the operation area is diminished and the amount of fat over device may be reduced to an extent that was unexpected at first implant. The change of device due to battery depletion can result in even less surrounding tissue. An alternative approach is an intramuscular placement of the device.7,8 This has been advocated by Kistler et al based on personal experience but there are neither systematic observational studies nor randomized controlled studies to support this approach.6 To the knowledge of the investigators no randomized controlled trial have addressed the question about the optimal placement of a bradycardia pacemaker.

Aim: To compare patient satisfaction with intramuscular placement of a pacemaker pocket to subcutaneous placement.

Research questions: Primary outcome: Is there a different in patient overall satisfaction (on a Visual Analog Scale (VAS)-scale between 0-10) with the pocket between patients with intramuscular placement of a pacemaker pocket and patients with subcutaneous placement at 24 months after implant? Secondary outcomes: Complications (revision of pocket, dislodgement, hematoma requiring surgery, infection (local/systemic). Patient reported satisfaction at 1, 12, 24 months (overall satisfaction, pain, discomfort, degree of unsightly look, movement problems due to device, and sleep problems due to device). Pacemaker nurse judgement of unsightly look of the pacemaker pocket (month 1, 12, and 24). Picture of pocket (1, 12, 24 months) judged by an experienced implanting physician who is blinded to the group allocation and has not operated on the patient.

Method: Power analysis: the investigators performed a power analysis based on expectations and clinical experience of the research group. Figure 1 shows two hypothetical truncated lognormal distributions of patient overall satisfaction with the pacemaker, where median overall satisfaction of the intramuscular and the subcutaneous group are assumed to be 2.4 and 4, respectively. Monte Carlo-simulations from these distributions showed that a total of 200 patients, 100 in each arm, would yield a statistical power of 90% for Mann-Whitney U-test at a significance level of 0.05.

In total, 200 consecutive patients with indication of are expected to be randomized in the study (100 patients in each arm, intramuscular vs subcutaneously). In Region Gavleborg , the annual primary implant volume of bradycardia pacemakers is approximately 220.

Figure 1. Assumed distributions of patient overall satisfaction in the power analysis, as measured by an visual analogue scale where 0 means "very satisfied" and 10 means "very dissatisfied". The intramuscular group is assumed to follow a lognormal distribution with mean 1.5 and standard deviation of 1, on the logarithmic scale. The subcutaneous patients are assumed to follow a lognormal distribution with mean 1.5 and standard deviation of 1, on the logarithmic scale.

Randomization: At the time of implant 1:1 randomization (100 patients in each group) to either subcutaneous (usual care) or intramuscular implant, in blocks with random block sizes. The randomization is performed by a statistician with no insight in the ongoing clinical work and patients' group allocation is revealed for implanting physician by the assistant nurse at the start of the surgical procedure. Randomization procedure: stratification (age strata: ≤65 years and >65 years) and sex (female, male); totally 4 strata). Consecutive group allocations will be stored in sealed opaque envelopes that will be opened at the time of starting the implant procedure.

Inclusion: Indication of a bradycardia pacemaker (DDDR, VVIR). Exclusion: Cardiac Resynchronisation Therapy Pacemaker (CRTP), Cardiac Resynchronisation Therapy Defibrillator (CRTD), implantable cardioverter defibrillator (ICD). Very skinny patient deemed as such by implanting physician to clearly benefit from intramuscular implant.

Surgical procedure: Standard procedure and vascular access by each operator's preference. Blunt dissection of the pocket.

Statistical methods: For comparisons between groups: Mann-Whitney U-test. For test of changes in VAS-estimations between 1, 12, and 24 months: pair-wise Wilcoxon signed-rank test.

Informed consent: Written and oral information by nurse/physician before implant.

Ethical approval: Approved by Uppsala Regional Committee. Clinical Trial Registration: Registration before start of study.

Variables:

Clinical variables: age, sex, coronary artery disease, open-heart surgery, diabetes, kidney disease Pacemaker system: (VVIR, DDDR), brand, model (lead(s) and device. Vascular access: (cephalic, axillary, subclavian vein), fluro-time, procedure time Periprocedural analgetics (dosage): alfentanil, morphine, diazepam, paracetamol Pre och post-operative anticoagulant medication (dosage and withdrawal with respect to procedure: acetylic acid, clopidogrel, ticagrelor, dual oral anticoagulants, warfarin, low-molecular weight heparin) Preoperative current medication: (psychoactive drugs, betablockers, corticosteroids, inflammatory modulating drugs Outcome measurements: Patient satisfaction (overall, chronic pain, discomfort, degree of unsightly look, movement disorder due to device, sleep problems due to device) scale 0-10 (10 worst) Paper questionnaire at 1,12,and 24 months. Patient knowledge if device was intramuscular or subcutaneously implanted at 24 months.

Pacemaker nurse judgement: unsightly look (0-10, 10 worst). Physician evaluation (blinded to the patient and not operator in the study): photo of pocket (1, 12, 24 months) scale 0-10 (10 worst).

Complications requiring surgery: pocket revision, dislodgment, hematoma requiring surgery, infection (local, systemic), pneumothorax, pericardial effusion requiring drainage, other.

Clinical perspectives: The surgical approach to the pacemaker pocket needs to be evaluated. The optimal approach including patient reported outcomes may result in more long-term satisfaction and may reduce the need for pocket revisions.

ELIGIBILITY:
Inclusion Criteria:

* Indication of a bradycardia pacemaker (DDDR, VVIR).

Exclusion Criteria:

* CRTP, CRTD, ICD.
* Very skinny patient deemed as such by implanting physician to clearly benefit from intramuscular implant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
patient overall satisfaction | 24 months
  Is there a different in patient overall satisfaction (on a VAS-scale between 0-10) with the pocket between patients with intramuscular placement of a pacemaker pocket and patients with subcutaneous placement at 24 months after implant?

SECONDARY OUTCOMES:
complications due to pacemaker procedure | 24 months
  Complications (revision of pocket, dislodgement, hematoma requiring surgery, infection (local/systemic). Measurement: number of each event (n)
pain problems due to pacemaker device | 24 months
  Patient reported pain at 1, 12 and 24 months on a VAS-scale 0-10.
discomfort due to pacemaker device | 24 months
  Patient reported discomfort at 1, 12, 24 months on a VAS-scale 0-10.
Patient own judgement of degree of unsightly look due to pacemaker device | 24 months
  Patient reported satisfaction at 1, 12, 24 months on a VAS-scale 0-10.
movement problems due to device | 24 months
  Patient reported satisfaction at 1, 12, 24 months on a VAS-scale 0-10.
sleep problems due to device | 24 months
  Patient reported satisfaction at 1, 12, 24 months on a VAS-scale 0-10.
Pacemaker nurse judgement of unsightly look of the pacemaker pocket | 24 months
  Pacemaker nurse judgement of unsightly look of the pacemaker pocket (month 1, 12, and 24) on a VAS-scale 0-10.
Picture of pocket | 24 months
  Picture of pocket (1, 12, 24 months) judged by an experienced implanting physician who is blinded to the group allocation and has not operated on the patient on a VAS-scale 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Per Liv, Ph.D, Principal Investigator — Centre for Research and Development Gavleborg/Uppsala University
Locations (1):
- Region Gavleborg, Gävle, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available (without identification of each individual) upon request by the journal (i.e Supplement file)

REFERENCES:
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822
- [Background] Gadler F, Valzania C, Linde C. Current use of implantable electrical devices in Sweden: data from the Swedish pacemaker and implantable cardioverter-defibrillator registry. Europace. 2015 Jan;17(1):69-77. doi: 10.1093/europace/euu233. Epub 2014 Oct 21. PMID 25336667
- [Background] Rajappan K. Permanent pacemaker implantation technique: part II. Heart. 2009 Feb;95(4):334-42. doi: 10.1136/hrt.2008.156372. No abstract available. PMID 19176569
- [Background] Rajappan K. Permanent pacemaker implantation technique: part I: arrhythmias. Heart. 2009 Mar;95(3):259-64. doi: 10.1136/hrt.2007.132753. No abstract available. PMID 19144885
- [Background] Kirkfeldt RE, Johansen JB, Nohr EA, Jorgensen OD, Nielsen JC. Complications after cardiac implantable electronic device implantations: an analysis of a complete, nationwide cohort in Denmark. Eur Heart J. 2014 May;35(18):1186-94. doi: 10.1093/eurheartj/eht511. Epub 2013 Dec 17. PMID 24347317
- [Background] Kistler PM, Fynn SP, Mond HG, Eizenberg N. The subpectoral pacemaker implant: it isn't what it seems! Pacing Clin Electrophysiol. 2004 Mar;27(3):361-4. doi: 10.1111/j.1540-8159.2004.00442.x. PMID 15009864
- [Background] Gold MR, Peters RW, Johnson JW, Shorofsky SR. Complications associated with pectoral implantation of cardioverter defibrillators. World-Wide Jewel Investigators. Pacing Clin Electrophysiol. 1997 Jan;20(1 Pt 2):208-11. doi: 10.1111/j.1540-8159.1997.tb04844.x. PMID 9121991